CLINICAL TRIAL: NCT04535375
Title: Sonographic Quantification of Venous Circulation in the Preterm Brain
Acronym: SQUIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Fleur Anne Camfferman, Principle investigator, Clinical professor, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SQUIB2020
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Prematurity; Extreme; Cerebral Circulatory Failure; Intraventricular Hemorrhage; Periventricular Leukomalacia
Keywords: Preterm infant, extremely preterm infant; Cerebral circulation; Venous Flow; Internal Cerebral Vein; Neurodevelopmental outcome; Intraventricular Hemorrhage; Periventricular Leukomalacia
MeSH Terms: conditions — Premature Birth; Leukomalacia, Periventricular

STUDY DESIGN:
Intervention Model Description: All stable preterm infants born before a gestational age of 32 weeks are eligible for inclusion.
  Since standard ultrasound protocol is different for preterm infants born below or after 28 weeks, two subgroups will be created.
Who Masked: Outcomes Assessor
Masking Description: Extra ultrasound images will be exported anonymized and analyses offline by two investigators independently
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preterm infants < 28 weeks gestational age (Other): For infants born before 28 0/7 weeks, standard of care consists of brain ultrasound performed on admission, day 1, day 2, day 3, day 7, and then weekly until discharge.
  Interventions: Diagnostic Test: Doppler Ultrasound of venous cerebral circulation
- Preterm infants born between 28 0/7 and 31 6/7 weeks (Other): For infants born between 28 0/7 and 31 6/7 weeks, brain ultrasound is performed on admission, once between day 1 and 3, once between day 7 and 10, and then 2-weekly until discharge or transfer.
  Interventions: Diagnostic Test: Doppler Ultrasound of venous cerebral circulation

INTERVENTIONS:
Diagnostic Test: Doppler Ultrasound of venous cerebral circulation — No additional ultrasound examinations, specifically for the purpose of this study, will be performed. Instead, with each routine ultrasound examination, additional images on top of the routine frames will be collected. Those images will document the velocity and flow in the internal cerebral veins bilaterally using the standard Color Doppler tech-nique. Taking these additional images will prolong the time of ultrasound examination only minimally (with a few minutes).

SUMMARY:
The aim of the study is to develop an accessible, reproducible ultrasound tool for objective clinical measurement of brain circulation in preterm infants in order to identify infants being at risk for preterm brain injury at an early stage. In the future, the results of this study might be useful to select those infants for early interventions aimed at preventing brain injury.

In this study we will identify the normative values of the internal cerebral vein velocity in a reference cohort of stable preterm infants. This stable group of preterm infants is defined as all preterm infants with a birth weight appropriate for gestational age, and without major complications (such as a severe intracranial hemorrhage, severe hemodynamical instability, birth asphyxia) or major congenital malformations.

In this group we will identify subgroups based on moments of clinical instability (sepsis, temporary hypotension, NEC, need for invasive respiratory support) or based on outcome parameters (IVH, PVL, developmental outcomes)

DETAILED DESCRIPTION:
The aim of the study is to develop an accessible, reproducible ultrasound tool for objective clinical measurement of brain circulation in preterm infants in order to identify infants being at risk for preterm brain injury at an early stage. In the future, the results of this study might be useful to select those infants for early interventions aimed at preventing brain injury.

In this study we will identify the normative values of the internal cerebral vein velocity in a reference cohort of stable preterm infants. This stable group of preterm infants is defined as all preterm infants with a birth weight appropriate for gestational age, and without major complications (such as a severe intracranial hemorrhage, severe hemodynamical instability, birth asphyxia) or major congenital malformations.

In this group we will identify subgroups based on moments of clinical instability (sepsis, temporary hypotension, NEC, need for invasive respiratory support) or based on outcome parameters (IVH, PVL, developmental outcomes)

Serial brain ultrasound examinations are routinely performed as standard of care after preterm birth for timely de-tection of brain hemorrhage in the first week of life and brain injury in the weeks thereafter until term equivalent age. For infants born between 28 0/7 and 31 6/7 weeks, brain ultrasound is performed on admission, once between day 1 and 3, once between day 7 and 10, and then 2-weekly until discharge or transfer. For infants born before 28 0/7 weeks, standard of care consists of brain ultrasound performed on admission, day 1, day 2, day 3, day 7, and then weekly until discharge.

No additional ultrasound examinations, specifically for the purpose of this study, will be performed. Instead, with each routine ultrasound examination, additional images on top of the routine frames will be collected. Those images will document the velocity and flow in the internal cerebral veins bilaterally using the standard Color Doppler tech-nique. Taking these additional images will prolong the time of ultrasound examination only minimally (with a few minutes).

The ultrasound will be performed using a standardized ultrasound protocol according to Ecury-Goossen et al (18) us-ing the Esaote MyLab Twice (Genova, Italy) with a linear (Esaote LA 435 Linear Array Ultrasound Probe, 6.0-18.0 MHz) and convex probe (Esaote CA123 Convex Array Ultrasound Probe, 3.3-9.0 MHz). This is the standard ultra-sound machine for ultrasound investigations at our neonatology ward.

For routine cranial ultrasound, ten images are generally made through the anterior fontanelle: five in the coronal and five in the sagittal plane. In addition to that, color Doppler or power Doppler is commonly performed in one of the pericallosal arteries in order to evaluate the arterial circulation, quantified by calculating a resistency index (RI). Usually routine ultrasound takes up to 10-15 minutes.

After routine scanning, four extra images will be acquired. These are power doppler images, one per insonated ves-sel of interest. The vessels of interest are the internal cerebral vein (left and right separate, if feasible) and one small tributary (the posterior caudate vein) on each side. To derive these images the duration of the US will be prolonged with approximately 3-5 minutes.

Blood flow velocities (maximum velocity and velocity pattern (17)) can be calculated offline in the anonymously ex-ported dicom file of these four images.

In addition to the ultrasound data, the following clinical patient data will be collected during the study:

* Data on systemic perfusion immediately before each ultrasound: arterial blood pressure, mixed cerebral oxygen saturation using near infrared spectroscopy (NIRS), fractional oxygen extraction, limb oxygen satu-ration, heart rate and use of inotropes.
* Demographic data during hospitalization, such as gender, gestational age, birth weight, head circumfer-ence and complications during hospitalization (infection, surgery, etcetera).

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant with a gestational age below 32 0/7 weeks
* birth weight between the 3rd and 97th percentile.
* No cerebral Doppler abnormalities on prenatal ultrasound (i.e. brain sparing)

Exclusion Criteria:

* Brain vessel anomaly
* Major congenital malformation
* No parental consent
* IVH > grade 2 (Papile classification or structural brain abnormalities on the first ultrasound
* Severe hemodynamic instability in the first 6 hours of life requiring treatment with inotropes.

Max Age: 3 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Normative values of internal cerebral vein velocity | 2-3 years
  Determination of normative values of ICV velocity and their range in the first weeks of life in stable preterm infants. The Doppler measurements will be performed at several moments after birth: day 0, 1, 2, 3, 7, 14, 21, etc untill 36 weeks gestational age.
  For this purpose we will calculate the Maximum velocity (cm/s), the mean velocity (cm/s) and the variability (according to Ikeda et al) of the flow pattern in the Internal Cerebral Vein. These velocities will be plotted in an attempt to discover longitudinal normative values in this cohort of 50 preterm infants.

SECONDARY OUTCOMES:
Short-term outcome: cerebral complications in the neonatal phase | 2-3 years
  Relation of ICV flow with IVH grade 2 or more (according to the Papile classification), periventricular leukomalacia, ventriculomegaly, white matter disease, selective neuronal necrosis assessed by routinely performed MRI scan of the brain at term equivalent age.
Long-term outcome: neurodevelopmental impairment | 3-5 years
  Relation of ICV flow with Bayley mental and motor scales at 2 years of age, as rou-tinely performed by the COS - Centrum voor Ontwikkelingsstoornissen.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Govaert, MD PhD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
For future systematic reviews anonimized individual participant data can be made available is an e-mail request is addressed at the principal investigator.

REFERENCES:
- [Background] Papile LA, Burstein J, Burstein R, Koffler H. Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm. J Pediatr. 1978 Apr;92(4):529-34. doi: 10.1016/s0022-3476(78)80282-0. PMID 305471
- [Background] Osborn DA, Evans N, Kluckow M. Hemodynamic and antecedent risk factors of early and late periventricular/intraventricular hemorrhage in premature infants. Pediatrics. 2003 Jul;112(1 Pt 1):33-9. doi: 10.1542/peds.112.1.33. PMID 12837865
- [Background] Kluckow M, Evans N. Low superior vena cava flow and intraventricular haemorrhage in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2000 May;82(3):F188-94. doi: 10.1136/fn.82.3.f188. PMID 10794784
- [Background] Caicedo A, Naulaers G, Lemmers P, van Bel F, Wolf M, Van Huffel S. Detection of cerebral autoregulation by near-infrared spectroscopy in neonates: performance analysis of measurement methods. J Biomed Opt. 2012 Nov;17(11):117003. doi: 10.1117/1.JBO.17.11.117003. PMID 23117814
- [Background] de Waal KA, Evans N, Osborn DA, Kluckow M. Cardiorespiratory effects of changes in end expiratory pressure in ventilated newborns. Arch Dis Child Fetal Neonatal Ed. 2007 Nov;92(6):F444-8. doi: 10.1136/adc.2006.103929. Epub 2007 Apr 25. PMID 17460022
- [Background] Hamon I, Hascoet JM, Debbiche A, Vert P. Effects of fentanyl administration on general and cerebral haemodynamics in sick newborn infants. Acta Paediatr. 1996 Mar;85(3):361-5. doi: 10.1111/j.1651-2227.1996.tb14033.x. PMID 8695997
- [Background] Skov L, Hellstrom-Westas L, Jacobsen T, Greisen G, Svenningsen NW. Acute changes in cerebral oxygenation and cerebral blood volume in preterm infants during surfactant treatment. Neuropediatrics. 1992 Jun;23(3):126-30. doi: 10.1055/s-2008-1071327. PMID 1641080
- [Background] Caicedo A, De Smet D, Naulaers G, Ameye L, Vanderhaegen J, Lemmers P, Van Bel F, Van Huffel S. Cerebral tissue oxygenation and regional oxygen saturation can be used to study cerebral autoregulation in prematurely born infants. Pediatr Res. 2011 Jun;69(6):548-53. doi: 10.1203/PDR.0b013e3182176d85. PMID 21364491
- [Background] van Bel F, Mintzer JP. Monitoring cerebral oxygenation of the immature brain: a neuroprotective strategy? Pediatr Res. 2018 Aug;84(2):159-164. doi: 10.1038/s41390-018-0026-8. Epub 2018 Aug 16. PMID 29907853
- [Background] Couture A, Veyrac C, Baud C, Saguintaah M, Ferran JL. Advanced cranial ultrasound: transfontanellar Doppler imaging in neonates. Eur Radiol. 2001;11(12):2399-410. doi: 10.1007/s00330-001-1150-z. Epub 2001 Oct 30. PMID 11734933
- [Background] Camfferman FA, de Goederen R, Govaert P, Dudink J, van Bel F, Pellicer A, Cools F; eurUS.brain group. Diagnostic and predictive value of Doppler ultrasound for evaluation of the brain circulation in preterm infants: a systematic review. Pediatr Res. 2020 Mar;87(Suppl 1):50-58. doi: 10.1038/s41390-020-0777-x. PMID 32218536
- [Background] Kluckow M, Evans N. Superior vena cava flow in newborn infants: a novel marker of systemic blood flow. Arch Dis Child Fetal Neonatal Ed. 2000 May;82(3):F182-7. doi: 10.1136/fn.82.3.f182. PMID 10794783
- [Background] Evans N, Kluckow M, Simmons M, Osborn D. Which to measure, systemic or organ blood flow? Middle cerebral artery and superior vena cava flow in very preterm infants. Arch Dis Child Fetal Neonatal Ed. 2002 Nov;87(3):F181-4. doi: 10.1136/fn.87.3.f181. PMID 12390987
- [Background] McGovern M, Miletin J. A review of superior vena cava flow measurement in the neonate by functional echocardiography. Acta Paediatr. 2017 Jan;106(1):22-29. doi: 10.1111/apa.13584. Epub 2016 Sep 28. PMID 27611695
- [Background] Lee A, Liestol K, Nestaas E, Brunvand L, Lindemann R, Fugelseth D. Superior vena cava flow: feasibility and reliability of the off-line analyses. Arch Dis Child Fetal Neonatal Ed. 2010 Mar;95(2):F121-5. doi: 10.1136/adc.2009.176883. Epub 2009 Dec 8. PMID 19996328
- [Background] Ikeda T, Amizuka T, Ito Y, Mikami R, Matsuo K, Kawamura N, Fusagawa S. Changes in the perfusion waveform of the internal cerebral vein and intraventricular hemorrhage in the acute management of extremely low-birth-weight infants. Eur J Pediatr. 2015 Mar;174(3):331-8. doi: 10.1007/s00431-014-2396-1. Epub 2014 Aug 30. PMID 25169064
- [Background] Ecury-Goossen GM, Camfferman FA, Leijser LM, Govaert P, Dudink J. State of the art cranial ultrasound imaging in neonates. J Vis Exp. 2015 Feb 2;(96):e52238. doi: 10.3791/52238. PMID 25742241
- [Background] Pfannschmidt J, Jorch G. Transfontanelle pulsed Doppler measurement of blood flow velocity in the internal jugular vein, straight sinus, and internal cerebral vein in preterm and term neonates. Ultrasound Med Biol. 1989;15(1):9-12. doi: 10.1016/0301-5629(89)90126-9. PMID 2646807
- [Background] Jansen-van der Weide MC, Caldwell PH, Young B, de Vries MC, Willems DL, Van't Hoff W, Woolfall K, van der Lee JH, Offringa M. Clinical Trial Decisions in Difficult Circumstances: Parental Consent Under Time Pressure. Pediatrics. 2015 Oct;136(4):e983-92. doi: 10.1542/peds.2014-3402. PMID 26416935
- [Background] Woolfall K, Frith L, Gamble C, Young B. How experience makes a difference: practitioners' views on the use of deferred consent in paediatric and neonatal emergency care trials. BMC Med Ethics. 2013 Nov 6;14:45. doi: 10.1186/1472-6939-14-45. PMID 24195717
- [Background] Woolfall K, Frith L, Gamble C, Gilbert R, Mok Q, Young B; CONNECT advisory group. How parents and practitioners experience research without prior consent (deferred consent) for emergency research involving children with life threatening conditions: a mixed method study. BMJ Open. 2015 Sep 18;5(9):e008522. doi: 10.1136/bmjopen-2015-008522. PMID 26384724